CLINICAL TRIAL: NCT03938818
Title: Targeted Interventions to Address the Multi-level Effects of Gender-based Violence on PrEP Uptake and Adherence Among Adolescent Girls and Young Women in Siaya County, Kenya
Brief Title: Tu'Washindi na PrEP: Adolescent Girls in Kenya Taking Control of Their Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Impact Research & Development Organization (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSU/DRPI/MUERC/00418/17; 1R34MH114519-01 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-05-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Gender-Based Violence
Keywords: Gender-Based Violence; PrEP (Pre-exposure Prophylaxis); AIDS Prevention; HIV Prevention

STUDY DESIGN:
Intervention Model Description: cluster randomized-controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard of care will include PrEP delivery according to the usual DREAMS procedures
  Interventions: Other: Control
- Tu'Washindi intervention (Experimental): Standard of care will include PrEP delivery according to the usual DREAMS procedures. The Tu'Washindi intervention includes the following components:
  1. PrEP sensitization for men (community level).
  2. "Buddy Days" (partner level).
  3. Adherence support clubs (individual and peer levels).
  Interventions: Behavioral: Tu'Washindi intervention

INTERVENTIONS:
Behavioral: Tu'Washindi intervention — The intervention includes the following components:
  1. PrEP sensitization for men (community level). These activities will aim to provide men with basic information about PrEP and will be used to prepare men for more effective engagement in Buddy Days, described below.
  2. "Buddy Days" (partner level). Buddy days will target male partner engagement by inviting couples to attend a community-wide event with health screenings, and PrEP sensitization, which aim to facilitate further communications about PrEP and increase men's support for AGYW's PrEP use.
  3. Adherence support clubs (individual and peer levels). Support clubs will provide a forum for AGYW to discuss challenges and successes around PrEP use in relationships, including in the context of partner violence. Participation in these groups is hypothesized to increase self-efficacy for PrEP use by reducing social isolation and providing additional positive role-modeling from peer leaders.
  Arms: Tu'Washindi intervention
Other: Control — Standard of care will include PrEP delivery according to the usual DREAMS procedures, including attendance at routine Safe Space meetings and routine PrEP provision at the Safe Space, if applicable.
  Arms: Control

SUMMARY:
This study is nested within the ongoing DREAMS (Determined, Resilient, Empowered, AIDS-free, and Safe) initiative in Siaya County, Kenya. It will test a pilot intervention that will address barriers to pre-exposure prophylaxis (PrEP) uptake and adherence in adolescent girls and young women (AGYW) to reduce their risk to HIV acquisition, with a focus on barriers stemming from male partners and gender-based violence.

DETAILED DESCRIPTION:
This study is designed to assess feasibility, safety, and preliminary effects of a behavioral intervention aimed at increasing pre-exposure prophylaxis (PrEP) uptake and adherence in adolescent girls and young women (AGYW), with a focus on barriers stemming from male partners and gender-based violence, through a pilot cluster randomized-controlled trial (RCT). This study is nested within the ongoing DREAMS (Determined, Resilient, Empowered, AIDS-free, and Safe) initiative in Siaya County, Kenya. Six DREAMS Safe Spaces and their catchment areas will be randomized to receive this community-level intervention or standard of care. Primary outcomes will include feasibility (recruitment, retention) and safety (ongoing or renewed experience of GBV). The investigators will also determine whether the intervention shows promise in increasing PrEP uptake, adherence, and persistence at 6 months. After the intervention, small group discussions, in-depth interviews with male partners, and provider questionnaires will explore acceptability and effects on PrEP decision making and use.

Population: AGYW ages 15-24 enrolled in the DREAMS Initiative in Siaya County, Kenya, and, for in-depth interviews only, a subset of male partners of DREAMS participants.

Objectives: The goal of this work is to test the feasibility, acceptability, safety, and preliminary effects of the intervention on PrEP uptake and adherence among AGYW.

The primary objectives are to assess:

1. Intervention safety
2. Feasibility of delivering the intervention within DREAMS operations
3. Acceptability of the intervention to participants, staff, and male partners.

The secondary objectives are to measure the intervention's effect on PrEP uptake, adherence, and persistence at 6 months.

Endpoints: The endpoints for the primary objectives are:

1. Self-report of new or ongoing GBV, social harms, serious adverse events, or unanticipated problems during study participation, in the intervention arm versus the comparison arm.
2. Measures of feasibility including recruitment, retention, intervention participation, and fidelity of intervention delivery.
3. Qualitative and quantitative reports of intervention acceptability among participants, quantitative reports of acceptability among providers, and qualitative reports of acceptability among male partners.

The endpoints for the secondary objectives are:

1. PrEP uptake: Among participants who are not on PrEP at study enrollment, the proportion of who receive a PrEP prescription during follow-up in the intervention arm vs. the control arm
2. PrEP adherence: Among participants who were dispensed PrEP during the study, the proportion with >85% adherence over the duration of PrEP use and in the last month of PrEP use, according to Wisepill data in the intervention arm vs. the control arm.
3. PrEP persistence: Among study participants who were dispensed PrEP during the study, the proportion of scheduled PrEP refills that were dispensed, in the intervention arm compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 15-24 years (inclusive);
* 2) HIV-negative, by self-report;
* 3) At high risk for acquiring HIV, as defined by the 2016 Guidelines on Use of Antiretroviral Drugs for Treating and Preventing HIV Infections in Kenya;
* 4) Fluent in English, Dholuo, or Swahili;
* 5) Enrolled in DREAMS (defined by having a DREAMS identification (ID) number);
* 6) Lives within the Safe Space catchment area - 7) Willing and able to attend support groups over the 6-month period;
* 8) Potentially interested in PrEP and/or using PrEP already;
* 9) Able and willing to provide adequate locator information, as defined in site standard operating procedures (SOPs);
* 10)If aged 18 and above: Willing and able to provide informed consent;
* 11)If non-mature minor aged 15-17: Willing and able to provide assent and parent or guardian willing and able to provide parental consent;
* 12)If mature minor aged 15-17: Willing and able to provide informed consent or to provide assent and parent or guardian consent, per participant choice.

Exclusion Criteria:

* 1)Planning to relocate away from the study catchment area in the next 6 months;
* 2)Planning to travel away from the study catchment area for a time period that would interfere with study participation; or
* 3) Has any condition that, in the opinion of the site PI, would preclude informed assent/consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Intervention safety - survey tool | 3 months
  Self-report of experience of social harms in the past 3 months and violence or controlling behavior using an adapted version of the World Health Organization's questions on violence against women. Behaviors are reported for every experience in the past 3 months and frequency of experience (e.g., once, few times, many times).
Intervention safety - survey tool | 6 months
  Self-report of experience of social harms in the past 3 months and violence or controlling behavior using an adapted version of the World Health Organization's questions on violence against women. Behaviors are reported for every experience in the past 3 months and frequency of experience (e.g., once, few times, many times).
Intervention safety - form | Throughout the study, approximately 6 months
  Reports of new or ongoing gender-based violence (GBV), social harms, serious adverse events, or unanticipated problems during study participation. Information will be self-reported using an specially-developed form
Feasibility of the behavioral intervention - Process Indicators | Throughout the study, approximately 6 months
  Measures of feasibility including recruitment timelines and numbers enrolled, retention rates, intervention participation measured by attendance at support club sessions and other intervention activities, and fidelity of intervention delivery measured through documented observations of intervention delivery capturing activities administered and ratings of quality.
Acceptability of the behavioral intervention - qualitative data from participants | 6 months
  Acceptability measures include qualitative reports of intervention acceptability among participants. These will include in-depth interviews covering topics such as satisfaction with content, delivery, and length of the intervention, as well as reported impact on the participant's life.
Acceptability of the behavioral intervention - quantitative data from participants | 6 months
  Quantitative reports of intervention acceptability among participants. Satisfaction with intervention content, delivery, length using the client satisfaction questionnaire and as measured on a likert scale response and as open-ended response options.
Acceptability of the behavioral intervention - quantitative data from providers | 6 months
  Satisfaction with intervention content, delivery, length using the client satisfaction questionnaire and as measured on a likert scale response and as open-ended response options.
Acceptability of the behavioral intervention - qualitative data from male partners | 6 months
  Qualitative reports of intervention acceptability among male partners. These will include in-depth interviews covering topics such as satisfaction with content, delivery, and length of the intervention, as well as reported impact on the male partner's life.

SECONDARY OUTCOMES:
Pre-Exposure Prophylaxis (PrEP) uptake | 6 months
  Among participants who are not on PrEP at study enrollment, the number who receive a PrEP prescription during follow-up. This will be measured through retrospective clinic record extraction.
Proportion of participants with Pre-Exposure Prophylaxis (PrEP) adherence > 85% at six months | Throughout the study, approximately 6 months
  Among participants who were dispensed PrEP during the study, the proportion with >85% adherence over the duration of PrEP use and in the last month of PrEP use, according to Wisepill data. This information will be collected using the Wisepill electronic data monitoring (EDM) device that collects information on pill adherence in real-time.
Pre-Exposure Prophylaxis (PrEP) persistence among participants at six months | 6 months
  Among study participants who were dispensed PrEP during the study, the number of scheduled PrEP refills that were dispensed. This will be measured through retrospective clinic record abstraction reflecting clinic visits throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Roberts, PhD, Principal Investigator — RTI International
Locations (1):
- Impact Research and Development Organization, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No